CLINICAL TRIAL: NCT04588311
Title: A Randomised, Double-blind, Placebo-controlled Trial of Erythropoietin Alfa Versus Placebo in Mechanically Ventilated Critically Ill Patients Following Traumatic Injury
Brief Title: ErythroPOietin Alfa to Prevent Mortality and Reduce Severe Disability in Critically Ill TRAUMA Patients
Acronym: EPO-TRAUMA
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Australian and New Zealand Intensive Care Research Centre (Other)
Collaborators: University College Dublin (Other); Medical Research Institute of New Zealand (Other); Medical Research Future Fund (Other); Health Research Board, Ireland (Other); Health Research Council, New Zealand (Other); Irish Critical Care Clinical Trials Network (Unknown); ANZICS Clinical Trials Group (Network); Monash University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ANZIC-RC/CF001; U1111-1242-3694 (Registry Identifier: Australian New Zealand Clinical Trials Registry (ANZCTR)); 2020-003388-24 (EudraCT Number)
Record Dates: First submitted 2020-10-01; First posted 2020-10-19 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Trauma; Traumatic Injury; Traumatic Brain Injury; Wounds and Injuries; Penetrating Injury; Blunt Injury; Major Trauma; Multiple Trauma
Keywords: Intensive Care Unit; Trauma; Major trauma; Traumatic injury; EPO; Erythropoietin; Epoetin alfa
MeSH Terms: conditions — Wounds and Injuries; Brain Injuries, Traumatic; Wounds, Penetrating; Wounds, Nonpenetrating; Multiple Trauma | interventions — Epoetin Alfa; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Erythropoietin (EPO) (Active Comparator): Epoetin alfa 40,000 IU (1mL pre-filled syringe) will be given by subcutaneous injection to eligible patients on Study Days 1 and 8 during the intensive care unit stay.
  Interventions: Drug: Epoetin Alfa 40000 UNT/ML
- Placebo (Placebo Comparator): Sodium Chloride 0.9% (1mL in volume) will be given by subcutaneous injection to eligible patients allocated to the placebo arm on Study Days 1 and 8 during the intensive care unit stay.
  Interventions: Drug: Sodium Chloride 0.9%

INTERVENTIONS:
Drug: Epoetin Alfa 40000 UNT/ML — Epoetin alfa 40,000IU 1mL pre-filled syringe given as subcutaneous injection.
  Other Names: Eprex; Binocrit
  Arms: Erythropoietin (EPO)
Drug: Sodium Chloride 0.9% — Sodium Chloride 0.9% 1mL in volume given as subcutaneous injection.
  Other Names: Placebo; Saline
  Arms: Placebo

SUMMARY:
The EPO-TRAUMA study is a prospective, multi-centre, double-blind, phase III, randomised controlled trial evaluating the efficacy of epoetin alfa compared to placebo in reducing mortality and severe disability at six months in critically ill trauma patients.

2500 mechanically ventilated ICU patients admitted with a primary trauma diagnosis presenting to the ICU will be recruited into the study from participating study centres in Australia, New Zealand, Europe, and Saudi Arabia.

DETAILED DESCRIPTION:
Trauma can cause many injuries, some of which are life-threatening and require treatment in an intensive care unit (ICU). Despite best available treatment and therapies, people who sustain a critical traumatic injury are at greater risk of death or long-term disability. From 2010 to 2015, approximately 9% of people admitted to an ICU in Australia and New Zealand for treatment of their injuries, did not survive. In Victoria, 6-months post injury, approximately 31% of people who were critically injured developed severe disabilities or died.

Following a traumatic injury, a number of complex pathways are activated by the body. These pathways can occur over hours or weeks and may lead to damage of cells, tissues or blood vessels and may destroy other healthy tissue. The treatment of traumatic injury focuses on trying to minimise further damage that can occur after the initial injury.

Erythropoietin is a glycoprotein hormone essential for erythropoiesis and was first purified in 1977. Its human recombinant analogues known as erythropoiesis stimulating agents (ESAs) are approved for human therapeutic use. However, erythropoietin is also a pleiotropic cytokine with effects beyond just erythropoiesis. Studies in animals have demonstrated the potential protective effects of erythropoietin to organs including the brain, kidney, liver and heart, and anti-inflammatory properties.

Previous research suggests the use of the ESA called epoetin alfa, increases the number of patients surviving severe trauma and reduces the risk of disability in those who survive.

The primary aim of the study is to determine the efficacy of epoetin alfa compared to placebo in reducing mortality and severe disability at six months in critically ill trauma patients.

2500 mechanically ventilated ICU patients admitted with a primary trauma diagnosis presenting to the ICU will be recruited into the study from participating study centres in Australia, New Zealand, Europe, and Saudi Arabia.

ELIGIBILITY:
Inclusion Criteria: Patients with trauma admitted to the ICU who:

* Are ≥ 18 to ≤ 75 years of age
* Are < 24 hours since primary traumatic injury
* Are invasively mechanically ventilated
* Are expected to stay in the ICU ≥ 48 hours
* Have a haemoglobin not exceeding the upper limit of the applicable normal (ULN) reference range in clinical use at the treating institution
* Have informed consent from a legal surrogate according to local law

Exclusion Criteria: Patients will be excluded from the study if any of the following criteria apply:

* GCS = 3 and fixed dilated pupils
* Recent history of DVT, PE or other thromboembolic event (within previous 12 months or receiving concomitant anticoagulant treatment for this indication)
* A chronic hypercoagulable disorder, including known malignancy
* Treatment with EPO in the last 30 days
* First dose of study drug unable to be given within 24 hours of primary injury
* Pregnancy or lactation or 3 months postpartum
* Expected to die imminently (< 24 hours)
* Known sensitivity to mammalian cell derived products
* Known contraindication to epoetin alfa
* End stage renal failure (receives chronic dialysis)
* Severe pre-existing physical or mental disability or severe co-morbidity that may interfere with the assessment of outcome
* The treating physician believes it is not in the best interest of the patient to be randomised to this trial

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2500 (Estimated)
Dates: Start 2020-11-09 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Combined proportion of participants who have died or have severe disability (WHODAS 2.0 > 25) | 6-months

SECONDARY OUTCOMES:
Mortality at 6-months | 6 months
Mortality at ICU discharge | 6-months
Mortality at Hospital discharge | 6-months
Mortality at day 28 | 28 days
Proportion of participants with a favourable Glasgow Outcome Score Extended (GOSE) (GOSE 5-8) compared to those have have died (GOSE 1), or have severe disability (GOSE 2-4). | 6-months
Proportion of participants with composite thrombotic vascular events (deep vein thrombosis (DVT), pulmonary embolism (PE), myocardial infarction (PI), cardiac arrest and cerebrovascular events) at 6 months. | 6-months

CONTACTS AND LOCATIONS:
Overall Officials: Associate Professor Craig French, Study Chair — Western Health; ANZIC Research Centre; Professor Alistair Nichol, Study Chair — University College Dublin
Locations (41):
- Australia (17):
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - St Vincent's Hospital Sydney, Darlinghurst, New South Wales
  - St George Hospital, Kogarah, New South Wales
  - Liverpool Hospital, Liverpool, New South Wales
  - John Hunter Hospital, New Lambton Heights, New South Wales
  - Royal North Shore Hospital, Saint Leonards, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Royal Darwin Hospital, Tiwi, Northern Territory
  - Cairns Hospital, Cairns, Queensland
  - Royal Brisbane and Women's Hospital, Herston, Queensland
  - Gold Coast University Hospital, Southport, Queensland
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Flinders Medical Centre, Adelaide, South Australia
  - The Alfred Hospital, Melbourne, Victoria
  - Royal Melbourne Hospital, Melbourne, Victoria
  - Royal Perth Hospital, Perth, Western Australia
- Belgium (6):
  - Cliniques Universitaires Saint-Luc, Brussels
  - HUB Hopital Erasme, Brussels
  - CHU-Charleroi Chimay, Charleroi
  - Ziekenhuis Oost-Limburg, Genk
  - Ghent University Hospital, Ghent
  - CHR de la Citadelle de LIEGE, Liège
- Finland (3):
  - Helsinki University Hospital (HUS), Helsinki
  - Kuopio University Hospital, Kuopio
  - Turku University Hospital, Turku
- University Hospital Münster, Münster, Germany
- Ireland (3):
  - Beaumont Hospital, Beaumont
  - Cork University Hospital, Cork
  - St Vincent's University Hospital, Dublin
- New Zealand (5):
  - Auckland City Hospital, Grafton, Auckland
  - Christchurch Hospital, Christchurch, Christchurch
  - Middlemore Hospital, Auckland, Otahuhu
  - Waikato Hospital, Hamilton, Waikato Region
  - Wellington Hospital, Newtown, Wellington Region
- King Abdulaziz Medical City, Riyadh, Saudi Arabia
- Slovenia (2):
  - University Medical Centre Ljubljana, Ljubljana
  - University Medical Centre Maribor, Maribor
- Switzerland (3):
  - University Hospital Bern, Bern
  - Lucerne Cantonal Hospital, Lucerne
  - St. Gallen Cantonal Hospital, Sankt Gallen

IPD SHARING:
Plan to Share IPD: Yes
At the conclusion of the study, the study management committee will consider requests from researchers who provide a methodically sound scientific proposal as per the Data Sharing Policy set out in the ANZIC-RC Terms of Reference.
Time Frame: As per the ANZIC Research Centre Data Sharing Policy
Access Criteria: As per the ANZIC Research Centre Data Sharing Policy

REFERENCES:
- [Background] Nichol A, French C, Little L, Haddad S, Presneill J, Arabi Y, Bailey M, Cooper DJ, Duranteau J, Huet O, Mak A, McArthur C, Pettila V, Skrifvars M, Vallance S, Varma D, Wills J, Bellomo R; EPO-TBI Investigators; ANZICS Clinical Trials Group. Erythropoietin in traumatic brain injury (EPO-TBI): a double-blind randomised controlled trial. Lancet. 2015 Dec 19;386(10012):2499-506. doi: 10.1016/S0140-6736(15)00386-4. Epub 2015 Oct 6. PMID 26452709